CLINICAL TRIAL: NCT05031546
Title: Intermediate-Size Patient Population Expanded Access Program for Intravenous Difelikefalin
Status: Approved for marketing | Type: Expanded Access
Sponsor: Cara Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CR845-500301
Record Dates: First submitted 2021-08-26; First posted 2021-09-02 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Uremic Pruritus
Keywords: Hemodialysis; Pruritus; Uremic Pruritus; Dialysis; CR845; Difelikefalin; Chronic Itch; CKD; CKD-associated pruritus; CKD-aP; ESRD (end stage renal disease); Itch; Itching; KALM; Chronic Kidney Disease; Kidney failure, chronic; Kidney dysfunction; Generalized pruritus; Expanded access; Compassionate use
MeSH Terms: conditions — Pruritus; Renal Insufficiency, Chronic; Kidney Failure, Chronic | interventions — difelikefalin

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: Difelikefalin — IV Difelikefalin 0.5 mcg/kg administered after each dialysis session (3 times/week)

SUMMARY:
This is an intermediate-size patient population expanded access protocol for the use of intravenous (IV) difelikefalin for the treatment of moderate-to-severe pruritus associated with chronic kidney disease in adult patients undergoing hemodialysis.

DETAILED DESCRIPTION:
Visits during the expanded access program will consist of a Baseline Visit to confirm eligibility and an End of Treatment visit. Patients will receive IV difelikefalin at a dose of 0.5 mcg/kg after each dialysis session, generally 3 times per week. The End of Treatment visit will be defined as the first dialysis visit following the last dose of IV difelikefalin under the intermediate-size patient population expanded access protocol.

ELIGIBILITY:
Key Inclusion Criteria:

* Adults ≥ 18 years old;
* Has end-stage renal disease (ESRD) and is currently receiving in-center hemodialysis;
* Has moderate-to-severe pruritus attributed to ESRD which is significantly impacting the patient's quality of life;
* Has no comparable or satisfactory alternative therapy for the treatment of moderate-to-severe pruritus, as determined by the sponsor-investigator.

Key Exclusion Criteria:

* Has severe hepatic impairment (Child-Pugh class C), as the influence of severe hepatic impairment on the pharmacokinetics of difelikefalin has not been evaluated;
* Is pregnant or nursing;
* Has been exposed to any other investigational medication in the past 60 days;
* Present any other reason which may lead to an unfavorable risk-benefit ratio for treatment with difelikefalin, as determined by the sponsor-investigator;
* Has a known or suspected allergy to difelikefalin or any component of the investigational product.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult